CLINICAL TRIAL: NCT04597372
Title: The Impact of Tamsulosin on Duration of Post-Operative Urinary Retention in Women Undergoing Pelvic Reconstructive Surgery- A Double Blind, Randomized, Placebo-Controlled Study
Brief Title: Impact of Tamsulosin on Post-Operative Urinary Retention Following Pelvic Reconstructive Surgery
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Lindsay Turner, Director of Urogynecology, Principal Investigator, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00264995
Record Dates: First submitted 2020-10-05; First posted 2020-10-22 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Urinary Retention Postoperative
MeSH Terms: interventions — Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tamsulosin (Experimental): 10 capsules will be distributed to subjects to be taken daily. Each capsule contains 0.4mg of Tamsulosin. Subjects will take the capsule once daily until the end of the 10 day course or until the resolution of acute postoperative urinary retention.
  Both study drug and placebo will appear identical and will be prepared by the pharmacy.
  Interventions: Drug: Tamsulosin
- Placebo (Placebo Comparator): 10 capsules will be distributed to subjects to be taken daily. Subjects will take the capsule once daily until the end of the 10 day course or until the resolution of acute postoperative urinary retention.
  Both study drug and placebo will appear identical and will be prepared by the pharmacy.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tamsulosin — Study drug will contain 0.4 mg of Tamsulosin. Subjects will be provided with 10 capsules to be taken daily.
  Arms: Tamsulosin
Drug: Placebo — Placebo will be prepared by the IDS pharmacist (or contracted pharmacy) and encapsulated in identical appearing wraps. Subjects will be provided with 10 capsules to be taken daily.
  Arms: Placebo

SUMMARY:
The objective of the study is to determine the effectiveness of postoperative Tamsulosin in reducing the duration of acute postoperative urinary retention (POUR) following pelvic reconstructive surgery through a double blind, randomized placebo-controlled trial.

DETAILED DESCRIPTION:
The primary objective is to determine the impact of Tamsulosin on duration of urinary retention following pelvic reconstructive surgery in women. Duration of catheterization via indwelling foley or clean intermittent self-catheterization (CISC), measured in days, will be compared between women receiving Tamsulosin versus placebo after diagnosis of postoperative urinary retention via standardized voiding trial. It is hypothesized that women receiving Tamsulosin will have a shorter duration of urinary retention, fewer urinary tract infections, and improved quality of life as compared with placebo. The Euroqol-5D (EQ-5D) will be used to compare physical, emotional, functional, and social/family well-being between women receiving Tamsulosin and placebo.

Upon diagnosis of POUR, women will be offered participation in the study. Once consent is obtained, women will be randomized to tamsulosin 0.4 mg or matching placebo capsules to be used daily until resolution of POUR or a 10 day course, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* willing and able to provide informed consent
* postoperative urinary retention as defined by a failed RGVT prior to hospital discharge
* Ability to speak and read English
* Tolerate pill ingestion

Exclusion Criteria:

* allergy/intolerance to Tamsulosin or sulfa drugs
* preoperative history of urinary retention as defined by preoperative post void residual of >150mL
* current use of alpha antagonist medication for hypertension
* severe dementia
* end stage renal or liver disease
* history of severe heart failure or major cardiovascular event in the last 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2021-11-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To determine the impact of Tamsulosin on duration of urinary retention | Date of failed retrograde voiding trial until resolution of post-operative urinary retention or a 10-day course
  The primary outcome is duration of postoperative urinary retention measured in days following failed retrograde voiding trial.

SECONDARY OUTCOMES:
To assess the impact of Tamsulosin on rates of urinary tract infection (UTI). | Date of failed the retrograde voiding trial and up to 6 weeks.
  The electronic medical record (EMR) will be reviewed to determine if subjects were treated for a urinary tract infection (UTI). UTIs will be diagnosed by a urine culture confirming bacteriuria of at least 10 ^5 CFU/mL. UTIs treated presumptively and without culture will also be included as positive cultures.
To quantify the effect of Tamsulosin on patient quality of life. | Prior to discharge and again at 2 weeks follow up
  Patients will be asked to complete the Euroqol-5D (EQ-5D) questionnaire to assess quality of life. The EQ-5D is scored with a 5-digit code of index values which reflect how good or bad a health state is (Level 1 indicates no problem where is Level 5 indicates extreme problems).

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Turner, MD, Principal Investigator — Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Locations (1):
- West Penn Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Results will be published; patient identifiers will not be used in the research publications.

REFERENCES:
- [Background] Willis-Gray MG, Wu JM, Field C, Pulliam S, Husk KE, Brueseke TJ, Geller EJ, Connolly A, Dieter AA. Is a Postvoid Residual Necessary? A Randomized Trial of Two Postoperative Voiding Protocols. Female Pelvic Med Reconstr Surg. 2021 Feb 1;27(2):e256-e260. doi: 10.1097/SPV.0000000000000743. PMID 31157716
- [Background] Geller EJ, Hankins KJ, Parnell BA, Robinson BL, Dunivan GC. Diagnostic accuracy of retrograde and spontaneous voiding trials for postoperative voiding dysfunction: a randomized controlled trial. Obstet Gynecol. 2011 Sep;118(3):637-642. doi: 10.1097/AOG.0b013e318229e8dd. PMID 21860294
- [Background] Oliphant SS, Lowder JL, Ghetti C, Zyczynski HM. Effect of a preoperative self-catheterization video on anxiety: a randomized controlled trial. Int Urogynecol J. 2013 Mar;24(3):419-24. doi: 10.1007/s00192-012-1868-y. Epub 2012 Jul 3. PMID 22752014
- [Background] Hooton TM, Bradley SF, Cardenas DD, Colgan R, Geerlings SE, Rice JC, Saint S, Schaeffer AJ, Tambayh PA, Tenke P, Nicolle LE; Infectious Diseases Society of America. Diagnosis, prevention, and treatment of catheter-associated urinary tract infection in adults: 2009 International Clinical Practice Guidelines from the Infectious Diseases Society of America. Clin Infect Dis. 2010 Mar 1;50(5):625-63. doi: 10.1086/650482. PMID 20175247
- [Background] K Ramakrishnan, J Mold. Urinary Catheters: A Review. The Internet Journal of Family Practice. 2004 Volume 3 Number 2.
- [Background] Baldini G, Bagry H, Aprikian A, Carli F. Postoperative urinary retention: anesthetic and perioperative considerations. Anesthesiology. 2009 May;110(5):1139-57. doi: 10.1097/ALN.0b013e31819f7aea. PMID 19352147
- [Background] Kuipers PW, Kamphuis ET, van Venrooij GE, van Roy JP, Ionescu TI, Knape JT, Kalkman CJ. Intrathecal opioids and lower urinary tract function: a urodynamic evaluation. Anesthesiology. 2004 Jun;100(6):1497-503. doi: 10.1097/00000542-200406000-00023. PMID 15166570
- [Background] Darrah DM, Griebling TL, Silverstein JH. Postoperative urinary retention. Anesthesiol Clin. 2009 Sep;27(3):465-84, table of contents. doi: 10.1016/j.anclin.2009.07.010. PMID 19825487
- [Background] Lose G, Lindholm P. Prophylactic phenoxybenzamine in the prevention of postoperative retention of urine after vaginal repair: a prospective randomized double-blind trial. Int J Gynaecol Obstet. 1985 Sep;23(4):315-20. doi: 10.1016/0020-7292(85)90026-8. PMID 2866119
- [Background] Livne PM, Kaplan B, Ovadia Y, Servadio C. Prevention of post-hysterectomy urinary retention by alpha-adrenergic blocker. Acta Obstet Gynecol Scand. 1983;62(4):337-40. doi: 10.3109/00016348309156234. PMID 6138916
- [Background] Roehrborn CG, Siami P, Barkin J, Damiao R, Major-Walker K, Morrill B, Montorsi F; CombAT Study Group. The effects of dutasteride, tamsulosin and combination therapy on lower urinary tract symptoms in men with benign prostatic hyperplasia and prostatic enlargement: 2-year results from the CombAT study. J Urol. 2008 Feb;179(2):616-21; discussion 621. doi: 10.1016/j.juro.2007.09.084. Epub 2007 Dec 21. PMID 18082216
- [Background] Lepor H. Phase III multicenter placebo-controlled study of tamsulosin in benign prostatic hyperplasia. Tamsulosin Investigator Group. Urology. 1998 Jun;51(6):892-900. doi: 10.1016/s0090-4295(98)00126-5. PMID 9609623
- [Background] FDA Prescription Drug Advisory Rule for Tamsulosin. NDA 020579.C.F.R. Accessed 4/3/20. https://www.accessdata.fda.gov/scripts/cder/daf/index.cfm?event=overview.process&varApplNo=020579
- [Background] Mohammadi-Fallah M, Hamedanchi S, Tayyebi-Azar A. Preventive effect of tamsulosin on postoperative urinary retention. Korean J Urol. 2012 Jun;53(6):419-23. doi: 10.4111/kju.2012.53.6.419. Epub 2012 Jun 19. PMID 22741052
- [Background] Narayan P, Tewari A. A second phase III multicenter placebo controlled study of 2 dosages of modified release tamsulosin in patients with symptoms of benign prostatic hyperplasia. United States 93-01 Study Group. J Urol. 1998 Nov;160(5):1701-6. PMID 9783935
- [Background] Madani AH, Aval HB, Mokhtari G, Nasseh H, Esmaeili S, Shakiba M, Shakiba RS, Seyed Damavand SM. Effectiveness of tamsulosin in prevention of post-operative urinary retention: a randomized double-blind placebo-controlled study. Int Braz J Urol. 2014 Jan-Feb;40(1):30-6. doi: 10.1590/S1677-5538.IBJU.2014.01.05. PMID 24642148
- [Background] Walters SJ, Brazier JE. Comparison of the minimally important difference for two health state utility measures: EQ-5D and SF-6D. Qual Life Res. 2005 Aug;14(6):1523-32. doi: 10.1007/s11136-004-7713-0. PMID 16110932
- [Background] Harvie HS, Honeycutt AA, Neuwahl SJ, Barber MD, Richter HE, Visco AG, Sung VW, Shepherd JP, Rogers RG, Jakus-Waldman S, Mazloomdoost D; NICHD Pelvic Floor Disorders Network. Responsiveness and minimally important difference of SF-6D and EQ-5D utility scores for the treatment of pelvic organ prolapse. Am J Obstet Gynecol. 2019 Mar;220(3):265.e1-265.e11. doi: 10.1016/j.ajog.2018.11.1094. Epub 2018 Nov 22. PMID 30471259
- [Background] Turner LC, Zyczynski HM, Shepherd JP. Intravenous Acetaminophen Before Pelvic Organ Prolapse Repair: A Randomized Controlled Trial. Obstet Gynecol. 2019 Mar;133(3):492-502. doi: 10.1097/AOG.0000000000003102. PMID 30741813
- [Background] Turner LC, Kantartzis K, Shepherd JP. Predictors of postoperative acute urinary retention in women undergoing minimally invasive sacral colpopexy. Female Pelvic Med Reconstr Surg. 2015 Jan-Feb;21(1):39-42. doi: 10.1097/SPV.0000000000000110. PMID 25185611
- [Background] Clinicaltrial.gov. Preoperative Tamsulosin to Prevent Postoperative Urinary Retention After Surgery For Pelvic Floor Disorders Accessed 4/3/20: https://clinicaltrials.gov/ct2/show/NCT04232683?term=tamsulosin&draw=2&rank=1